CLINICAL TRIAL: NCT07030920
Title: Reducing Systemic Inflammation in People on Antiretroviral Therapy
Acronym: RESTART
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other); Clinique du Quartier Latin (Network); BC Women's Hospital & Health Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MP-02-2025-12725; II2-195573 (Other Grant/Funding Number: Canadian Institutes of Heallth Research)
Record Dates: First submitted 2025-06-05; First posted 2025-06-22 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Human Immunodeficiency Virus (HIV); Cardiovascular Risk Factor
Keywords: Fostemsavir; Rukobia; sgp120; Perivascular fat attenuation index (P-FAI); uncalcified plaque volume; Systemic inflammation; Cardiovascular Risk Factor
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — fostemsavir

STUDY DESIGN:
Intervention Model Description: Randomization will be done in a 1:1 ratio, with allocation in parallel arms, stratified by sex and participant statin use at recruitment, through a computerized algorithm with permuted blocks of randomly varying size, to ensure allocation concealment.
Who Masked: Outcomes Assessor
Masking Description: This trial will be conducted as an open-label study; however, assessors of the primary outcome (based on two CCTA scans) and of the biobank analyses will remain blinded to treatment allocation, as well as statisticians.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rukobia 600 mg daily (Experimental)
  Interventions: Drug: Fostemsavir
- Standard of care (SOC) (No Intervention): Participants will continue to follow their current ART regimen, as well as other medications prescribed by their treating physician throughout the trial

INTERVENTIONS:
Drug: Fostemsavir — Addition of fostemsavir to the patient's current antiretroviral regimen: once daily oral administration (Rukobia 600 mg extended-release tablets) for 24 months
  Arms: Rukobia 600 mg daily

SUMMARY:
This randomized, open-label clinical trial will evaluate whether adding fostemsavir to current antiretroviral therapy can reduce the risk of cardiovascular disease in people with well-controlled HIV. Researchers will compare imaging, clinical and biomarker outcomes between participants who receive fostemsavir in addition to their existing treatment and those who continue with standard care alone.

DETAILED DESCRIPTION:
A randomized, controlled trial of fostemsavir versus standard of care to curb comorbidity in people with well-controlled HIV. (Phase IIb study)

Background and hypothesis: People living with HIV, even when treated with antiretrovirals, develop early onset comorbidities such as cardiovascular disease, cognitive decline and frailty. In a subset of those, this could be due to residual viral particles driving chronic inflammation. Soluble glycoprotein 120 (sgp120) is detectable in close to a third of people living with HIV with undetectable HIV plasma viral loads. It is associated to increased inflammation and immune dysfunction.

People living with HIV with undetectable viral load but detectable soluble HIV gp120 (sgp120) are exposed to chronic inflammation, sustained immune dysfunction, and increased risk of comorbidity. The investigators hypothesize that the addition of fostemsavir, which has been shown to prevents the binding of sgp120 to the human CD4 receptor, to reduce cytokine burst and antibody-dependant cellular citotoxicity, decreased inflammation and immune dysfunction, leading to improved health.

Study population: People living with HIV on antiretroviral therapy, with undetectable viral load and detectable plasmatic sgp120.

Study intervention: The intervention will be either the addition of fostemsavir (Rukobia 600 mg daily) for 24 months to the patient's current ART regimen, or standard of care, which includes the continuation of the ARV regimen and other medications prescribed by their physicians.

Randomization: This is a randomized, open label study with blind outcome adjudication. Randomization will be done in a 1:1 ratio with allocation in parallel arms, stratified by sex and participant statin use at recruitment, through a computerized algorithm with permuted blocks of randomly varying size, to ensure allocation concealment.

Treatment groups:

Arm 1 (active):

* Once daily oral administration (600 mg extended-release tablet) for 24 months Arm 2 (Standard of care)
* Participants will continue to follow their current ART regimen, as well as other medications prescribed by their treating physician throughout the trial

Study procedures: At baseline, participants will undergo a CCTA, grip strenght, a B-CAM (online cognitive testing) and contribute blood to the study biobank. Participants will be randomized during the baseline visit, and those randomized to fostemsavir will start taking study treatment. Visits will be done at month 1, 6, 12, 18, 24 and 27. The duration of treatment will be 24 months. At month 24, the CCTA, grip strenght and cognition measures will be repeated. Participants will contribute to the biobank at each study visit.

Study outcomes:

Primary Outcome: Change in total uncalcified plaque volume between baseline and month 24, contrasted between fostemsavir and standard of care.

Imaging Secondary Outcome: Perivascular fat attenuation index at month 24, adjusted for baseline values.

Clinical Secondary Outcome: Clinical events - time to major adverse cardiovascular event, B-CAM (cognition testing) and grip strength at month 24 (adjusted for baseline values).

Biomarker Secondary Outcomes: Biomarkers identified in biobanking samples (virology, immunology, inflammation).

Safety Secondary Outcomes: Risk of adverse events and incidence of treatment discontinuation due to side effects.

A biomarker interim analysis will be performed when 50% of the planned samples size will have completed 1 year of follow-up. Pre-specified biomarker outcomes will be measured using the study-associated biobank.

The intervention will be either the addition of fostemsavir (Rukobia 600 mg daily) to the patient's current ART regimen, or the participant receiving the standard of care.

Statistical considerations:

The planned sample size is 150 (approxiimately 75 per arrm. ) Statistical analysis will be conducted by CITADEL (CRCHUM) after the closing of the study database, according to the statistical analysis plan, which will be registered before the analysis is conducted. All analyses will be done by intention-to-treat; patients will be analyzed in the group they were randomized to. Biobank analyses planned after 50% of participants completed the 12 months biobanking will be done by CITADEL after this part of the data collection is closed.

ELIGIBILITY:
Inclusion Criteria:

* 40 years or older, or have lived with HIV for 25 years or more, any sex;
* Undetectable HIV viral load (defined as last viral load measurement less than 50 copies/ml within the last 6 months);
* Presence of at least one cardiovascular risk factor among the following: longstanding HIV infection (25 years or more), hypertension, diabetes, past or present smoking, dyslipidemia, family history of early onset CVD in a first-degree relative (defined as younger than 55 in males or younger than 65 in females (80)), known previous cardiovascular disease (defined as past myocardial infarction, coronary revascularization, stroke, or coronary artery atherosclerosis with >= 50% stenosis demonstrated on coronary angiography or CCTA);
* Participants with past cardiovascular disease must be in a stable clinical condition as judged by the study clinicians;
* Past cardiovascular events are defined as having occurred at least 3 months before screening;
* Evidence of detectable plasmatic sgp120 levels at any point in the past year, using the assay described priorly and performed at CRCHUM in Dr Andrés Finzi's laboratory.

Exclusion Criteria:

* Known allergy to study drug;
* Concomitant treatment with strong cytochrome P450 (CYP3A) inducers, including but not limited to: carbamazepine, phenytoin (anticonvulsants), mitotane (antineoplastic), enzalutamide (androgen receptor inhibitor), rifampicin (antimycobacterial) and St John's wort (Hypericum perforatum, herbal supplement);
* Planning to become pregnant, pregnant, or breastfeeding (as requested per product monography (55)). Females of childbearing potential must have a negative pregnancy test at baseline visit, and follow contraception requirements throughout the treatment;
* Contraindication for CT scan use (estimated glomerular filtration rate [eGFR] less than 40ml/min using the Modification of Diet in Renal Diseases [MDRD] formula or iodine allergy);
* Elevated risk of prior ionizing radiation exposure outside clinical care exceeding 10 mSV over 3 years, per the investigator's judgement (eg. a participant with occupational ionizing radiation exposure, prior participation in clinical trials with multiple CT scans)
* Confirmed uncorrected QT value >500ms or confirmed QTcF >470 msec for women and >450 msec for men;
* Acquired/ congenital long QT syndrome;
* Current or anticipated treatment with any of the following medications: amiodarone, disopyramide, dofetilide, ibutilide, procainamide, sotalol, and quinidine;
* Unstable liver disease (as defined by any of the following: presence of ascites, encephalopathy, coagulopathy (INR > 2.0), hypoalbuminemia (<30 mg/ml), untreated esophageal or gastric varices, or persistently elevated bilirubinemia (>1.5x upper limit of normal [ULN]), known biliary abnormalities (except Gilbert's syndrome or asymptomatic gallstones or otherwise stable chronic liver disease per investigator assessment);
* ALT >=5 times the ULN, OR ALT >=3xULN and bilirubin >=1.5xULN with >35% direct bilirubin;
* History of liver cirrhosis with CHILD-PUGH classification C;
* Inability to provide informed consent;
* Life expectancy of less than 36 months;
* Inability to present to study visits;
* Participation in another interventional trial;
* Known Congestive heart failure with NYHA class 3 or 4.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-09-30 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Change in total uncalcified plaque volume between baseline and month 24 | From baseline to end of treatment (+ 24 months)
  The change in total uncalcified plaque volume between baseline and month 24 will be measured by coronary compted tomography angiography and contrasted between fostemsavir and standard of care

SECONDARY OUTCOMES:
Imaging outcome: Perivascular fat attenuation index at month 24, adjusted for baseline values | From baseline to end of treatment (+ 24 months)
  The perivascular fat attenuation index at month 24, adjusted for baseline values, will be measured by CCTA and contrasted between fostemsavir and standard of care
Time to Major Adverse cardiovascular Event (MACE) | From baseline to post-treatment visit (+ 27 months)
  The time to MACE will be recorded throughout the study. MACEs are defined as myocardial infarction, coronary revascularization by percutaneous coronary intervention or surgery, peripheral artery revascularization, stroke, hospitalization for heart failure or unstable angina, or cardiovascular death
Risk of severe and serious adverse events | From baseline to post-treatment visit (+ 27 months)
Grip strength at 24 months, adjusted for baseline | From baseline to end of treatment (+ 24 months)
  Grip strength, a marker of sarcopenia, will be measured at month 24, adjusted for baseline. Grip strength will be measured using the standard operating procedures common to the Canadian HIV and Aging Cohort Study (CHACS) and Women's Interagency HIV Study (WHIS).
Brief Cognitive Ability Measure (B-CAM) scores at month 24, adjusted for baseline | From baseline to end of treatment (+ 24 months)
  B-CAM scores will be measured at month 24, adjusted for baseline. B-CAM scores will be measured using a web-based measurement tool that has been developed for cognitive assessment in PWH. It can be administered in less than 30 minutes, has been shown to be superior to the Montreal Cognitive Assessment Score (MoCA) to assess cognition in PWH, and remains valid when used repetitively in the same individual, with no need to adjust for practice effects.

OTHER OUTCOMES:
Biological biomarkers of inflammation and immune dysfunction | From screening (up to T0 - 6 months) to post-treatment visit (T0 + 27 months)
  The analysis of biomarkers will be presented as evolution over time between the study groups.
  Following marker groups will be assessed:
  Biomarkers of systemic inflammation and biomarkers associated to CVD Immuno-serology Presence of HIV soluble gp120 Plasma fostemsavir concentration

CONTACTS AND LOCATIONS:
Overall Officials: Madeleine Durand, MD MSc FRCPC, Principal Investigator — CR CHUM
Locations (1):
- CR CHUM, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benlarbi M, Richard J, Bourassa C, Tolbert WD, Chartrand-Lefebvre C, Gendron-Lepage G, Sylla M, El-Far M, Messier-Peet M, Guertin C, Turcotte I, Fromentin R, Verly MM, Prevost J, Clark A, Mothes W, Kaufmann DE, Maldarelli F, Chomont N, Begin P, Tremblay C, Baril JG, Trottier B, Trottier S, Duerr R, Pazgier M, Durand M, Finzi A. Plasma Human Immunodeficiency Virus 1 Soluble Glycoprotein 120 Association With Correlates of Immune Dysfunction and Inflammation in Antiretroviral Therapy-Treated Individuals With Undetectable Viremia. J Infect Dis. 2024 Mar 14;229(3):763-774. doi: 10.1093/infdis/jiad503. PMID 38035854
- [Background] Richard J, Prevost J, Bourassa C, Brassard N, Boutin M, Benlarbi M, Goyette G, Medjahed H, Gendron-Lepage G, Gaudette F, Chen HC, Tolbert WD, Smith AB 3rd, Pazgier M, Dube M, Clark A, Mothes W, Kaufmann DE, Finzi A. Temsavir blocks the immunomodulatory activities of HIV-1 soluble gp120. Cell Chem Biol. 2023 May 18;30(5):540-552.e6. doi: 10.1016/j.chembiol.2023.03.003. Epub 2023 Mar 22. PMID 36958337
- [Background] Durand M, Sheehy O, Baril JG, Lelorier J, Tremblay CL. Association between HIV infection, antiretroviral therapy, and risk of acute myocardial infarction: a cohort and nested case-control study using Quebec's public health insurance database. J Acquir Immune Defic Syndr. 2011 Jul 1;57(3):245-53. doi: 10.1097/QAI.0b013e31821d33a5. PMID 21499115
- [Background] Durand M, Chartrand-Lefebvre C, Baril JG, Trottier S, Trottier B, Harris M, Walmsley S, Conway B, Wong A, Routy JP, Kovacs C, MacPherson PA, Monteith KM, Mansour S, Thanassoulis G, Abrahamowicz M, Zhu Z, Tsoukas C, Ancuta P, Bernard N, Tremblay CL; investigators of the Canadian HIV and Aging Cohort Study. The Canadian HIV and aging cohort study - determinants of increased risk of cardio-vascular diseases in HIV-infected individuals: rationale and study protocol. BMC Infect Dis. 2017 Sep 11;17(1):611. doi: 10.1186/s12879-017-2692-2. PMID 28893184